CLINICAL TRIAL: NCT06795308
Title: The Effect of Position on Pain, Bleeding, Hematoma and Vital Signs After Transfemoral Coronary Angiography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Mizgin Bakır, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MERSİNU2024-TFCA
Record Dates: First submitted 2024-12-05; First posted 2025-01-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Coronary Disease; Angiography
Keywords: position; transfemoral coronary angiography; pain; bleeding; hematoma
MeSH Terms: conditions — Coronary Disease; Pain; Hemorrhage; Hematoma

STUDY DESIGN:
Intervention Model Description: The first group will remain in the supine position for 6 hours after the Angiography procedure, and the treated leg will be kept straight and immobile. Patients will not move their legs during this period. A sandbag weighing approximately 4 kg will be placed over the catheter dressing for 6 hours to prevent bleeding and subcutaneous blood accumulation. For the first two hours, the patient will lie on his back and on a flat surface with his legs extended straight. During the remaining 4 hours, researchers will monitor the patient's bed head by raising it 15 degrees intermittently under the supervision of the doctor, and at the end of the 6th hour, the sandbag on the leg will be removed. Blood pressure, pulse rate, respiratory rate, body temperature, as well as pain level will be measured every two hours. In the second group, only the patient's bed head will remain flat and will not be elevated.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENTERPRISE GROUP (Active Comparator): The first group will remain in the supine position for 6 hours after the Angiography procedure, and the treated leg will be kept straight and immobile. Patients will not move their legs during this period. A sandbag weighing approximately 4 kg will be placed over the catheter dressing for 6 hours to prevent bleeding and subcutaneous blood accumulation. For the first two hours, the patient will lie on his back and on a flat surface with his legs extended straight. During the remaining 4 hours, investigators will monitor the patient's bed head by raising it 15 degrees intermittently under the supervision of the doctor, and at the end of the 6th hour, the sandbag on the leg will be removed. Blood pressure, pulse rate, respiratory rate, body temperature, as well as pain level will be measured every two hours.
  Interventions: Other: Bed Position and Head Elevation
- CONTROL GROUP (No Intervention): After the angiography procedure, the patient will remain in the supine position for 6 hours and the treated leg will remain straight and motionless. investigators will ask patients not to move their legs during this time. A sandbag weighing approximately 4 kg will be placed over the catheter dressing for 6 hours to prevent bleeding and subcutaneous blood accumulation. Patients will lie on their back and on a flat surface with their legs extended straight for 6 hours. At the end of the 6th hour, the sandbag on the leg is removed. Blood pressure, pulse rate, respiratory rate, body temperature, as well as pain level will be measured every 2 hours.

INTERVENTIONS:
Other: Bed Position and Head Elevation — The first group will remain in the supine position for 6 hours after the Angiography procedure, and the treated leg will be kept straight and immobile. Patients will not move their legs during this period. A sandbag weighing approximately 4 kg will be placed over the catheter dressing for 6 hours to prevent bleeding and subcutaneous blood accumulation. For the first two hours, the patient will lie on his back and on a flat surface with his legs extended straight. During the remaining 4 hours, investigators will monitor the patient's bed head by raising it 15 degrees intermittently under the supervision of the doctor, and at the end of the 6th hour, the sandbag on the leg will be removed. Blood pressure, pulse rate, respiratory rate, body temperature, as well as pain level will be measured every two hours.
  Arms: ENTERPRISE GROUP

SUMMARY:
In this study, it was aimed to determine the effect of the special position given to the patient after transfemoral coronary angiography (supine position that varies depending on the angles) on pain, bleeding, hematoma and vital signs.

DETAILED DESCRIPTION:
Since coronary angiography is an invasive procedure, the prevention of complications is critical for nursing care. As a result of this procedure, complications such as bleeding, local vascular problems such as hematoma, ecchymosis, pseudoaneurysm, pain and vasovagal reactions triggered by pain may occur. However, it is possible to minimize these complications with appropriate nursing approaches and care. By carefully monitoring patients before and after the procedure, nurses play an important role in reducing the risk of complications and ensuring patient safety.

The mobility of patients both in bed and in the room after coronary angiography may increase the rate of complications such as bleeding, pain and hematoma. For this reason, complete bed rest is traditionally recommended in addition to manual pressure application to stop bleeding after intervention in the femoral artery procedure. However, this approach may cause problems in terms of patient comfort and increases the workload of healthcare personnel. Sandbags are used to make prints in some clinics. However, while these bags cause pain and discomfort to patients due to lying still for a long time, they can also cause bleeding and hematoma due to slipping of the sandbag, and can be especially challenging for elderly patients. In this case, the methods that can be applied should be applied in a short time and easily. Positioning increases blood circulation and prevents contraction and spasm of the muscles. It is also easy and quick to apply. As a result of this method, the level of pain decreases. Positioning is effective in acute pain. It is not recommended to give a position without evaluating the general condition of the patient. An assessment of the overall situation is necessary to understand all of the patient's health needs and provide comprehensive care. This assessment helps to determine the patient's general health status, current symptoms, and needs. Positioning is also part of this assessment. The decrease in pain depending on the position reduces the patient's desire to move. This makes it easier to evaluate the patient in terms of the amount of bleeding and the risk of hematoma formation. In the literature, there are studies evaluating pain or hematoma after transfemoral coronary angiography by applying different methods. There is a study evaluating the effect of supine position on pain and hematoma. However, there are no studies evaluating the effect of four parameters including pain, bleeding, hematoma and vital signs. In order to eliminate this deficiency in the literature, it was aimed to evaluate the effect of supine position, which varies depending on the angles after transfemoral coronary angiography, on pain, bleeding amount, hematoma and vital signs in the patient. Four different hypothesis sets were established in the research. These; First Hypothesis Team H0: The position applied to transfemoral coronary angiography patients has no effect on pain.

H1: The position applied to transfemoral coronary angiography patients has an effect on pain.

Second Hypothesis Team H0: The position applied to transfemoral coronary angiography patients has no effect on bleeding.

H1: The position applied to transfemoral coronary angiography patients has an effect on bleeding.

Third Hypothesis Team H0: The position applied to transfemoral coronary angiography patients has no effect on hematoma formation.

H1: The position applied to transfemoral coronary angiography patients has an effect on hematoma formation.

Fourth Hypothesis Team H0: The position applied to transfemoral coronary angiography patients has no effect on vital signs.

H1: The position applied to transfemoral coronary angiography patients has an effect on vital signs Flow Process of the Study First Stage (Preparatory Stage): Appropriate environment arrangements will be made for the patients included in the intervention and control groups.

Second Phase (Implementation Phase): This phase will consist of ten steps. First step: In the first step of the application, patients who have undergone transfemoral coronary angiography in the Cardiology Service of Adana City Training and Research Hospital, who meet the research criteria and who are willing to participate in the research, will be given brief information about the research, and the "Informed Consent Form" will be filled out, and the written consent of the patients will be obtained.

Second step: Sample selection will be made in accordance with the inclusion, exclusion and exclusion criteria of the research, then randomization will be performed and two randomized groups will be formed. Patients will be informed about the purpose of the research and the research process, and the "Patient Introduction Form" will be filled, and the vital signs of the patients who will be in the intervention and control groups will be measured and recorded in the "Vital Signs Evaluation Form". According to the VAS, general body pain will be evaluated and recorded. Routine nursing care procedures will be applied to both groups. Patients will be followed up in the service until and after the transfemoral coronary angiography procedure.

Third step: In the transfemoral coronary angiography procedure; Before the angiography catheter is withdrawn after the trasnfemoral coronary angiography procedure of the patient in the intervention group and control group, the procedure area will be evaluated and recorded in terms of pain intensity, amount of bleeding and hematoma measure. The angiography catheter will be removed by the doctor.

Fourth step: At the 0th hour after transfemoral coronary angiography catheter is withdrawn; In the intervention group, the patient's bedhead 0 degree will be placed in the supine position with the treated leg straight and immobile, and in the control group, the patient's bedside 0 degree will be brought to the supine position with the treated leg straight and immobile, and a sandbag weighing 4 kg will be placed on the treated area. The patient will be evaluated for pain severity and vital signs will be measured and recorded.

Fifth step: At the 1st hour after the transfemoral coronary angiography catheter is removed; In the intervention group, the patient's bedhead 0 degree will be placed in the supine position with the treated leg straight and immobile, and in the control group, the patient's bedside 0 degree will be brought to the supine position with the treated leg straight and immobile, and a sandbag weighing 4 kg will be placed on the treated area.

Sixth step: Transfemoral coronary angiography at the 2nd hour after the catheter is removed; In the intervention group, the patient's bedside will be 15 degree, the treated leg will be placed in the supine position with straight and immobile, and in the control group, the patient's bedside will be 0 degree, the treated leg will be placed in the supine position with the treated leg straight and immobile, and a sandbag weighing 4 kg will be placed in the treated area. The patient will be evaluated in terms of pain severity, vital signs will be measured and recorded.

Seventh step: At the 3rd hour after the transfemoral coronary angiography catheter is withdrawn; In the intervention group, the patient's bedside will be 15 degree, the treated leg will be straight and immobile, and in the control group, the patient will be placed in a supine position with the patient's bedside 0 degree and the treated leg will be straight and immobile, and a sandbag weighing 4 kg will be placed on the treated area.

Eighth step: At the 4th hour after the transfemoral coronary angiography catheter is removed; In the intervention group, the patient's bedhead will be 30 degree, the treated leg will be placed in the supine position with the treated leg straight and immobile, and in the control group, the patient will be placed in the supine position with the patient's bedhead 0 degree and the treated leg straight and immobile, and a sandbag weighing 4 kg will be placed on the treated area. The patient will be evaluated in terms of pain severity, vital signs will be measured and recorded.

Ninth step: At the 5th hour after the transfemoral coronary angiography catheter is withdrawn; In the intervention group, the patient's bedside will be 45 degree, the treated leg will be placed in the supine position with the treated leg straight and immobile, and in the control group, the patient will be placed in the supine position with the patient's bedside 0 degree and the treated leg straight and immobile, and a sandbag weighing 4 kg will be placed in the treated area.

Tenth step: At the 6th hour after the transfemoral coronary angiography catheter is removed; The 4 kg sandbag of the patient in the intervention group and the control group will be removed. The patient's procedure area will be evaluated in terms of the amount of bleeding, hematoma size and pain severity, and vital signs will be measured and recorded.

Third Stage (Reporting Stage): At this stage, statistical analysis of the data obtained from the patients will be made and a research report will be written.

ELIGIBILITY:
Inclusion Criteria:

* Written and verbal permission was obtained to participate in the research.
* Able to read, write, speak and understand Turkish
* Those who are over 18 years old
* Planned transfemoral angiography was performed
* Having normal prothrombin time (PT) and international normalization ratio (INR)
* Being conscious, fully oriented and cooperative, and open to communication.
* Those whose general condition is good and comfortable (vital signs are within normal limits)
* Not using any sedative medication,
* Those who have not previously had widespread hemorrhage, large hematoma, or a pain sensation greater than 4.5 on the visual pain scale
* Patients with imaging, medical treatment, stents, balloons, stents and balloons as a result of the procedure
* Not having any psychiatric disease

Exclusion Criteria:

Exclusion criteria;

* People with hemophilia or other coagulation defects
* Those with active hemorrhage
* Previously treated with streptokinase
* Using more than 2 anticoagulants or antiplatelets
* Those who have had back surgery/herniated disc,
* Having chronic waist, back or leg pain
* Using any of the complementary and integrated methods
* Do not use any analgesic before, during and after transfemoral angiography.
* Radial angiography procedure was performed
* Patients coming to the service with sandbags
* Those who had any health problems or lost their lives during the application process
* Those who cannot continue the research for any reason
* Patients who wish to leave the study with their own consent

Min Age: 18 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women/men
Enrollment: 60 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Pre-intervention and after the intervention 6 hour.
  First evaluation criterion after transfemoral coronary angiography is pain. The results will be evaluated using the Visual Analog Scale. "No pain" is rated as 0 points (minimum value) and "very severe pain" is rated as 10 points (maximum value). Pain will decrease as Visual Analog Scale score decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Digdem LAFCI BAKAR, PhD, Principal Investigator — Mersin University
Locations (1):
- Adana City Training and Research Hospital, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 1 year after the publication date and without an end date
Access Criteria: Who Can Access: Access will only be open to analyzes by independent experts, academic institutions or approved health administrations. Access pieces will be evaluated as an independent review monitoring committee will evaluate them.
  What Will Be Accessed: Individual data (IPD) of the participants, the data in which they are presented, usage information (samples, analysis methods, data collection tools, etc.) will be shared.
  How They Will Access: Access may be removed through an application process that is maintained or accepted by the administrator. Once the request is approved and the application is approved, it will be accessed via special data access platforms or secure data storage areas.
  Types of Analysis: Sharing of data is only for analysis after an independent review committee has evaluated it. These analyzes need to be monitored, monitored, and analysis types need to be combined and committees created.

REFERENCES:
- [Result] Valiee S, Fathi M, Hadizade N, Roshani D, Mahmoodi P. Evaluation of feasibility and safety of changing body position after transfemoral angiography: A randomized clinical trial. J Vasc Nurs. 2016 Sep;34(3):106-15. doi: 10.1016/j.jvn.2016.05.001. PMID 27568318
- See also: PubMed — https://pubmed.ncbi.nlm.nih.gov/27568318/